CLINICAL TRIAL: NCT06485206
Title: A Clinical Investigation Evaluating Safety and Effectiveness of Primary Hybrid Construct of Mobi-C and ACDF in the Treatment of Two-level Symptomatic Degenerative Disc Disease in the Cervical Spine.
Brief Title: Evaluation of Safety and Effectiveness of Primary Hybrid Construct of Mobi-C and ACDF in the Treatment of Two-level Symptomatic Degenerative Disc Disease in the Cervical Spine.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Highridge Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Highridge Medical
Record Dates: First submitted 2024-06-19; First posted 2024-07-03 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-09

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Primary Hybrid Construct (Experimental): Primary hybrid surgery is when patients undergo CDA and ACDF at the same time.
  Interventions: Device: One level Mobi-C and one level fusion

INTERVENTIONS:
Device: One level Mobi-C and one level fusion — Cervical Disc Arthroplasty:
  • Mobi-C
  Fusion devices:
  * One-level cervical plates
    o MaxAn Cervical plate system
  * Interbody spacers
    * TrellOss-C - 3D printed Ti interbody
    * Vista-S - PEEK interbody
  * Standalone Fixation
    * Ti-Coated ROI-C - PEEK cage w/ Ti coating
    * TrellOss-C SA - 3D printed Ti
  * Bone Graft
    * Local Autograft
    * PrimaGen Advanced Allograft
  Other Names: Mobi-C Hybrid

SUMMARY:
The study is a prospective, multi-center cohort study of patients with two-level DDD implanted with CDA adjacent to ACDF (hybrid construct). The overall success of the hybrid procedure will be compared to 2-level ACDF historical controls from the Mobi-C IDE trial. 97 patients will receive the hybrid surgery and will be followed for a minimum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 22 - 69 years. 2. Have symptoms of cervical degenerative disc disease (DDD) at two levels from C3 to T1 defined as intractable radiculopathy (arm pain and /or a neurological deficit) with or without neck pain or myelopathy due to a two-level abnormality localized to the level of the disc space.

  3. Radiographic evidence of at least one of the following:

  a. Spondylosis (defined by the presence of osteophytes or dark disc) on CT or MRI; or b. Disc height decreased by ≥1 mm when compared to adjacent levels on radiographic film, CT, or MRI; or c. Disc herniation on CT or MRI. Appropriate treatment for using an anterior surgical approach, including having no prior surgery at the operative levels and no prior cervical fusion or arthroplasty procedure.

  4. Neck Disability Index Score of ≥15/50 or ≥30%. 5. Unresponsive to non-operative, conservative treatment (rest, heat, electrotherapy, physical therapy, chiropractic care and analgesics) for:
  1. Approximately six weeks from radiculopathy or myeloradiculopathy symptom onset; or
  2. Have the presence of progressive symptoms or signs of nerve root/spinal cord compression despite continued non-operative conservative treatment.

     6. Able and willing to comply with the Protocol, including ability to read and complete required forms and willing and able to adhere to the scheduled follow-up visits* and requirements of the Protocol 7. Written informed consent provided by subject or subject's legally authorized representative.

     *Note that patients who live significant distances away from a treatment center are statistically likely to be present for treatment but are not likely to return for all follow-up visits. For this reason, patients who live over 150 miles from a treatment center are not eligible for treatment in this clinical study without prior approval from the study Sponsor.

     Exclusion Criteria:
* 1. Symptomatic DDD or significant cervical spondylosis at more than two levels 2. Reported to have an active systemic infection or infection at the operative site 3. Previous trauma resulting in significant bony or disco-ligamentous cervical spine injury 4. More than one immobile vertebral level between C1 to C7 from any cause including but not limited to congenital abnormalities and osteoarthritic "spontaneous" fusions 5. Reported to have had any prior fusion or CDA surgery in the cervical spine 6. Axial neck pain only (no radicular or myelopathy symptoms) 7. Disc height ≤25% of the anterior-posterior width of the inferior vertebral body 8. Severe facet joint disease or degeneration; or evidence of symptomatic moderate to severe facet joint degeneration or disease where the investigator feels this is a major contributor to the patient's pain as diagnosed by injection and imaging 9. Marked cervical instability on resting lateral or flexion/extension radiographs demonstrated by:

  * Translation greater than 3.5mm, and/or
  * Greater than 11° angular difference to that of either adjacent level 10. Segmental angulation of greater than 11° at treatment or adjacent levels 11. Metabolic bone disease (e.g., osteoporosis/osteopenia, gout, osteomalacia, Paget's disease) 12. Reported to have osteoporosis (T-SCORE greater than -1.0). All patients 50 years and older, post-menstrual, and females with hysterectomies will undergo a DEXA scan or hologic sahara as part of the study enrollment procedures.
  * For patients less than 50 years of age, the Simple Calculated Osteoporosis Risk Estimation (SCORE) questionnaire will be used to screen patients for osteoporosis. Patients whose screening suggests risk will undergo a DEXA scan.
  * Patients will be excluded if the DEXA scan results indicate a T-SCORE worse than -1.0 13. Any disease, condition or surgery which might impair healing, such as: Diabetes mellitus requiring daily insulin management 14. Active malignancy 15. Known sensitivity or allergies to any of the materials used with any of devices in study (e.g., cobalt chromium, titanium, polyethylene, PEEK) 16. Reported pregnancy or nursing at time of enrollment 17. Reported to have rheumatoid arthritis, lupus, or other autoimmune disease that affect the musculoskeletal system 18. Congenital bony and/or spinal cord abnormalities that affect spinal stability 19. Reported to have diseases or conditions that would preclude accurate clinical evaluation (e.g. neuromuscular disorders) 20. Reported concomitant conditions requiring steroid treatment 21. Reported to be taking medications known to potentially interfere with bone/soft tissue healing, e.g., long term use of corticosteroids (this does not include inhalation medications for asthma) 22. Reported to have a current history of heavy smoking (no less than one pack of cigarettes per day) 23. Recent history (within previous six months) of chemical or alcohol dependence 24. Morbid obesity, as defined by NIH Clinical Guidelines Body Mass Index (BMI > 35) 25. Participation in any other investigational drug, biologic, or medical device study within the last 30 days prior to study surgery 26. Currently involved in spinal litigation or receiving Worker's Compensation related to neck or back pain which may influence the subjects reporting of symptoms 27. Reported to have mental illness or belongs to a vulnerable population as determined by the investigator (e.g., prisoner or developmentally disabled) that would compromise ability to provide informed consent or compliance with follow-up requirements 28. Reported to have an uncontrolled seizure disorder

Ages: 22 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Composite Success | 24 months
  Statistical analysis of the combination of four components of success: improvement in Neck Disability Scale scores, no device failures, no major complications resulting in reoperations, no major AEs

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | 24 months
  The Neck Disability Index (NDI) is a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain.
Visual Analogue Scale- Neck Pain | 24 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain in the neck.
Visual Analogue Scale- Arm Pain | 24 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain in the arms.
Muscle Strength | 24 months
  Clinical outcome
Sensory Deficit | 24 months
  An assessment made by the surgeon with a neurological examination to determine if there is any change in sensation compared to the assessment before surgery.
Neurological Deficit | 24 months
  An assessment made by the surgeon with a neurological examination to determine if there is any change in neurological function compared to the assessment before surgery.
Adjacent Segment Degeneration | 24 months
  Radiological assessment using Kellgren-Lawrence classification system to measure degeneration occurring in levels around the operated spine.
Heterotopic Ossification | 24 months
  Radiological assessment using McAfee to measure bony growth on areas of motion in the Mobi-C level of the operated spine.
Subsidence | 24 months
  Radiographic outcome
Segmental Range of Motion | 24 months
  Radiographic outcome
C2-C7 range of motion | 24 months
  radiographic outcome
radiolucency measure | 24 months
  radiographic outcome
Patient Satisfaction Questionnaire | 24 months
  Self-reported questionnaire to assess patient satisfaction of the surgical treatment outcomes
quality of life survey (SF-12) | 24 months
  Patient reported outcome measure
Dysphagia | 24 months
  Dysphagia will be assessed using Functional Outcome Swallowing Scale (FOSS)
Gait Analysis | 24 months
  Gait will be assessed by physician during neurological examination

OTHER OUTCOMES:
Duration of Hospitalization | 6 weeks
  Clinical outcome
Blood Loss | 6 weeks
  clinical outcome
Operative Time | intraoperative
  clinical outcome
Return to Work | 6 weeks
  Clinical outcome will be measured by patient self-report of time since surgery before returning to work measured in days.
Headache Outcome (HIT-6) | 24 months
  patient reported outcome

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California-Davis, Sacramento, California
  - Michigan Orthopaedic Surgeons, Southfield, Michigan

IPD SHARING:
Plan to Share IPD: No